CLINICAL TRIAL: NCT01092767
Title: Evaluation of the Clinical Performance of the Valiant Thoracic Stent Graft With the Captivia Delivery System for the Endovascular Treatment of Blunt Thoracic Aortic Injuries (RESCUE)
Brief Title: Study to Determine if the Valiant Stent Graft is Safe and Effective in Treating Patients Who Have a Blunt Thoracic Aortic Injury
Acronym: RESCUE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiovascular (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Investigational Plan #117
Record Dates: First submitted 2010-03-16; First posted 2010-03-25 (Estimated); Results first posted 2014-03-28 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Blunt Thoracic Aortic Injury
Keywords: Thoracic Aneurysm; Thoracic Transection; Endovascular Aortic Repair
MeSH Terms: conditions — Aortic Aneurysm, Thoracic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Valiant Thoracic Stent Graft with the Captivia Delivery System (Experimental): Valiant Thoracic Stent Graft with the Captivia Delivery System
  Interventions: Device: Valiant Thoracic Stent Graft with the Captivia Delivery System

INTERVENTIONS:
Device: Valiant Thoracic Stent Graft with the Captivia Delivery System — All subjects will be implanted with this device

SUMMARY:
The purpose of this study is to determine if the Valiant stent graft is safe and effective in treating patients who have a blunt thoracic aortic injury (BTAI). BTAI is when the aorta has been injured due to traumatic force to the chest area. It is commonly caused by motor vehicle accidents. In most cases it is life threatening and the standard treatment is surgery. Many times when a person has a BTAI they also have other injuries that can affect the results of the surgery.

Since stent grafting has been an effective way to treat other aortic conditions such as aneurysms (bulge in aorta wall), it is believed that the Valiant stent graft would be effective in treating BTAI. A stent graft is a woven polyester tube (graft) supported by a metal frame of strong but flexible nitinol (type of metal) springs (stent) that is placed in the aorta to help seal the injury and keep it from bleeding.

ELIGIBILITY:
Inclusion Criteria

* Subject had a blunt thoracic aortic injury which:
* was confirmed, at a minimum, by diagnostic contrast-enhanced computerized tomography angiogram (CTA) and/or contrast-enhanced magnetic resonance angiogram (MRA)
* occurred no more than 30 days prior to the stent implant procedure
* Subject was ≥ 18 years of age
* Subject or subject's legally authorized representative signed an IRB approved informed consent
* Subject was hemodynamically stable
* Subject's anatomy met all of the following anatomical criteria:
* Aortic diameter (adventitia to adventitia) of the proximal and distal landing zones between 18 mm and 44 mm
* Subject had patent iliac or femoral arteries or could tolerate an iliac conduit that allowed endovascular access to the injury site with the delivery system of the appropriate sized device
* The centerline distance from the distal margin of left common carotid artery (LCC) to the injury was ≥ 20 mm

Exclusion Criteria

* Planned placement of the COVERED portion of the stent graft over the celiac axis or the LCC, or in cases of bovine anatomy, innominate artery
* Subject had systemic infection
* Subject was pregnant
* Subject had received a previous stent or stent graft or previous surgical repair in the DTA
* Subject had a history of bleeding diathesis, coagulopathy, or refuses blood transfusion
* Subject was participating in an investigational drug or device clinical trial which would interfere with the endpoints and/or follow-ups of this study
* Subject had a known allergy or intolerance to the device components
* Subject had a known hypersensitivity or contraindication to anticoagulants or contrast media, which was not amenable to pre-treatment
* Subject was in extremis, defined as subject that had non-survivable injury/condition
* Subject had a Cerebral Vascular Accident (CVA) within two (2) months prior to implant procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2012-04 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodney White, MD, FACS, Principal Investigator — Harbor UCLA
Locations (25):
- United States (23):
  - University of Alabama, Birmingham, Alabama
  - Cedars Sinai Medical Center, Los Angeles, California
  - Harbor UCLA, Torrance, California
  - Denver Health, Denver, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - University of Florida Shands Hospital, Gainesville, Florida
  - University of Miami Jackson Memorial, Miami, Florida
  - Bayfront Medical Center, St. Petersburg, Florida
  - Maine Medical Center, Portland, Maine
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Cooper Health, Camden, New Jersey
  - Vascular Research Institute, Morristown, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - Toledo Hospital / Jobst Vascular Center, Toledo, Ohio
  - UT Southwestern, Dallas, Texas
  - Memorial Hermann Heart and Vascular Institute, Houston, Texas
  - Brooke Army Medical Center, San Antonio, Texas
  - Scott and White Memorial, Temple, Texas
  - University Of Virginia, Charlottesville, Virginia
  - Sentara Norfolk General Vascular & Transplant Specialists, Norfolk, Virginia
  - Medical College of Wisconsin Froedtert Hospital, Milwaukee, Wisconsin
- Canada (2):
  - London Health Sciences Center, London, Ontario
  - Laval Hospital, Québec

REFERENCES:
- [Derived] Khoynezhad A, Donayre CE, Azizzadeh A, White R; RESCUE investigators. One-year results of thoracic endovascular aortic repair for blunt thoracic aortic injury (RESCUE trial). J Thorac Cardiovasc Surg. 2015 Jan;149(1):155-61.e4. doi: 10.1016/j.jtcvs.2014.09.026. Epub 2014 Sep 19. PMID 25439771
- [Derived] Khoynezhad A, Azizzadeh A, Donayre CE, Matsumoto A, Velazquez O, White R; RESCUE investigators. Results of a multicenter, prospective trial of thoracic endovascular aortic repair for blunt thoracic aortic injury (RESCUE trial). J Vasc Surg. 2013 Apr;57(4):899-905.e1. doi: 10.1016/j.jvs.2012.10.099. Epub 2013 Feb 4. PMID 23384495

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 25 investigational sites were activated and allowed to enroll in the RESCUE study in the US and Canada. A total of 50 subjects were enrolled at 20 of the 25 activated investigational sites, with the first enrollment on April 14, 2010 and the final enrollment on January 17, 2012.
Pre-assignment Details: All 50 subjects enrolled were implanted with the device (Valiant Thoracic Stent Graft with the Captivia Delivery System ).
Groups:
- Valiant Thoracic Stent Graft With the Captivia Delivery System: Valiant Thoracic Stent Graft with the Captivia Delivery System : All subjects will be implanted with this device
Period: Overall Study
Arm/Group | Valiant Thoracic Stent Graft With the Captivia Delivery System
Started | 50
Completed | 45
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Valiant Thoracic Stent Graft With the Captivia Delivery System
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 43
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (17.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 38
Region of Enrollment [Number; unit: participants]
  United States | 48
  Canada | 2

OUTCOME MEASURES:

1. Primary Outcome: All-cause Mortality Within 30-days of the Index Procedure
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | Valiant Thoracic Stent Graft With the Captivia Delivery System
Number analyzed (Participants) | 50
participants | 4

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- 1. Rescue: Rescue
Arm/Group | 1. Rescue
Serious Adverse Events (participants affected / at risk) | 8/50
Other Adverse Events (participants affected / at risk) | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1. Rescue (N=50)
Arrhythmia (Cardiac disorders) | 1 (1)
Infection (Infections and infestations) | 0 (0)
Multiple Injuries (Injury, poisoning and procedural complications) | 1 (1)
Traumatic Brain Injury (Injury, poisoning and procedural complications) | 1 (1)
Anoxic Encephalopathy (Nervous system disorders) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Femoral Artery Dissection (Vascular disorders) | 1 (1)
Intermittent Claudication (Vascular disorders) | 1 (1)
Peripheral Ischaemia (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator (PI) and institution agree not to publish the results of the study until after the earliest of the following: a)conclusion of the study, b)the early termination of the study, c)at discretion and approval of the sponsor, or d)after sponsor confirms there will be no multicenter study publication, whichever occurs first. PI and institution further agree to submit to sponsor copies of any proposed publication or public presentation at least sixty days before dissemination.